CLINICAL TRIAL: NCT04630600
Title: Effect of the Presence of an Aquarium in the Waiting Room on the Pre-treatment Stress and Anxiety Levels of Adult Patients and Reception Staff: a Controlled Clinical Trial
Brief Title: Presence of Aquarium in the Waiting Room of a Geriatric Dental Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Murali Srinivasan, Professor, University of Zurich
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UZH_ABS_2020_1
Record Dates: First submitted 2020-11-03; First posted 2020-11-16 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Stress; Anxiety; Mood
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): Normal waiting room
  Interventions: Other: No intervention
- Intervention#1 (Experimental): Waiting room with partially-equipped aquarium (without fish)
  Interventions: Other: Partially-equipped aquarium in the waiting area
- Intervention#2 (Experimental): Waiting room with fully-equipped aquarium (with fish)
  Interventions: Other: Fully-equipped aquarium in the waiting area

INTERVENTIONS:
Other: No intervention — Normal waiting room without an aquarium
  Arms: Control
Other: Partially-equipped aquarium in the waiting area — Waiting room with a partially-equipped Aquarium
  Arms: Intervention#1
Other: Fully-equipped aquarium in the waiting area — Waiting room with a fully-equipped Aquarium
  Arms: Intervention#2

SUMMARY:
The participants in this study will be subjected to a specific clinic waiting area ambience (1- no aquarium, 2- presence of aquarium with no fish, and 3- aquarium with fish) for their period of waiting before their intended dental visit and their stress and anxiety levels will be measured. Heart rate, blood pressure will be measured and other upon their arrival into the dental clinic waiting area and then again after 20 minutes of waiting in the waiting area. Anxiety will be measured using a six-item State-Trait Anxiety Inventory (STAI-6) questionnaire and the mood of the participants were assessed for valence and arousal, using the feeling scale, and the felt arousal scale. The data from the three different waiting room settings will be compared and statistically analysed to investigate if an aquarium has an impact, and in that case how.

DETAILED DESCRIPTION:
Dental anxiety is a well-known, common dilemma affecting many adults, observed more frequently in children and women. It is an emotional apprehensive state which is multifactorial and the origin is most commonly attributed to the anticipation of the painful stimulus that may arise during treatment. It has been suggested that environmental factors contribute to dental stress. Although quite trivial, the environment of a waiting room as well as the time spent waiting are parameters that can cause pre- treatment stress. Therefore, the waiting room must be considered an important first port for dealing with the individual's pre-treatment dental anxiety. Evidence in literature suggest that waiting room ambience plays a significant role in reducing the patient anxiety, for example images, audio-visual effects like the lighting, music and/or videos, presence of natural light, suitable reading material, aquariums have shown positive results. Beneficial effects of the presence of animals on the reduction of stress have also been reported in literature, and especially fish have shown a positive effect on the psychological well-being and stress levels; higher relaxation, less anxiety and better mood was reported by participants after a period of observing live fish.

* The primary null hypothesis is that there will be no effect of an aquarium present in the waiting area on the pre-treatment anxiety and stress levels of participants receiving dental care.
* The secondary hypothesis is that there will be no effect of an aquarium present in the waiting area on the stress and anxiety levels of the reception staff.
* The tertiary hypothesis for this study is that the treating dentist will not perceive any difference in the stress and anxiety levels of the participants after observing the aquarium in the waiting area.
* Patients ≥18 years, who are able to sign a consent form are included. The participants are subjected to a specific clinic waiting area ambience (1- no aquarium, 2- presence of aquarium with no fish, and 3- aquarium with fish) for their period of waiting before their intended dental visit and their stress and anxiety levels are measured. Heart rate, blood pressure will be measured and other upon their arrival into the dental clinic waiting area. Three measurements will be taken and then after 20 minutes of waiting another three measurements of the same will be made in order to see if the presence of an aquarium gave a decrease. Anxiety will be measured using a six-item State-Trait Anxiety Inventory (STAI-6) questionnaire and the mood of the participants were assessed for valence and arousal, using the feeling scale, and the felt arousal scale. The data from the three different settings will be compared and statistically analysed to investigate if an aquarium has an impact, and in that case how.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Able to give informed consent as documented by signature.

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Visually impaired.
* Participants enrolled already in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure (systolic and diastolic) | Day 0
  Stress levels
Heart rate | Day 0
  Stress levels
STAI-6 | Day 0
  6-item Short State Trait Anxiety Inventory
Feeling scale | Day 0
  Mood
Felt Arousal Scale | Day 0
  Mood

CONTACTS AND LOCATIONS:
Overall Officials: Murali Srinivasan, Principal Investigator — University of Zurich
Locations (1):
- Clinic of General, Special care, and Geriatric Dentistry, Center of Dental Medicine, University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No